CLINICAL TRIAL: NCT05765500
Title: RecoverPC: A Phase 2 Study of RElugolix Versus GnRH Agonist Quality of Life (QOL) and Testosterone reCOVERy in Men With Prostate Cancer
Brief Title: RecoverPC: Relugolix vs GnRH Agonist in Quality of Life
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Prostate Cancer Foundation (Other); Pfizer (Industry); Myovant Sciences GmbH (Industry)
Responsible Party: Principal Investigator, Alicia Morgans, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-599
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
Keywords: Prostate Cancer; Prostate Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix; Leuprolide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Relugolix (Experimental): 55 participants will be randomized in a 1:1 fashion to Relugolix and stratified by intent to treat with radiation and will complete study procedures as outlined:
  * Surveys at baseline and at months 3, 6, 9, and 12.
  * Medication diary entries.
  * Cycles 1 - 6:
    --Days 1 - 28 of 28 day cycle: Predetermined dose of Relugolix. Participant will self-administer at home.
  * Follow up visits every 3 months for 12 months.
  Interventions: Drug: Relugolix
- Arm B: Leuprolide (Active Comparator): 55 participants will be randomized in a 1:1 fashion to Leuprolide and stratified by intent to treat with radiation and will complete study procedures as outlined:
  * Surveys at baseline and at months 3, 6, 9, and 12.
  * Cycle 1 and Cycle 4:
    --Day 1 of 28 day cycle: Predetermined dose of Leuprolide. Injection will be administered in clinic.
  * Follow up visits every 3 months for 12 months.
  Interventions: Drug: Leuprolide

INTERVENTIONS:
Drug: Relugolix — Gonadotropin-releasing hormone (GnRH) antagonist, oral tablet taken 1x daily.
  Other Names: Orgovyx
  Arms: Arm A: Relugolix
Drug: Leuprolide — Gonadotropin-releasing hormone (GnRH) antagonist, intramuscular injection 1x every 3 months.
  Other Names: Leuprolide Depot
  Arms: Arm B: Leuprolide

SUMMARY:
This study is testing the way that approved androgen deprivation therapy treatments, Leuprolide and Relugolix, for prostate cancer affect quality of life, blood levels, cholesterol, and blood sugar. The drugs are already standard treatment for people with prostate cancer, and the drugs will be used as described in their label.

The names of the study drugs involved in this study are:

* Leuprolide (type of ADT)
* Relugolix (type of ADT)

DETAILED DESCRIPTION:
This is a phase 2 clinical trial comparing patient-reported Quality of Life (QOL) among men with localized or biochemically recurrent prostate cancer treated with relugolix versus leuprolide depot therapy.

Participants will be randomized into one of the study groups leuprolide versus relugolix. Randomization means that a participant is put into a study group by chance.

The U.S. Food and Drug Administration (FDA) has approved leuprolide and relugolix as treatment options for prostate cancer.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits, ECGs, and blood tests.

Participation in this research study is expected to last 12 months.

It is expected about 110 people will take part in this research study.

The Prostate Cancer Foundation and Pfizer are supporting this research study by providing funding. Myovant is supporting this study by providing the drug, Relugolix.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologic diagnosis of prostate adenocarcinoma.
* Participants must be eligible for treatment with 6 months of ADT with leuprolide depot or relugolix without additional systemic therapies other than first generation androgen receptor antagonists (eg. bicalutamide, nilutamide, flutamide).
* Participants cannot have received prior GnRH agonist or antagonist therapy.
* Patients must have testosterone level > 200 ng/mL prior to initiation of ADT.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Life expectancy of greater than 12 months
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ institutional upper limit of normal (ULN) unless known or suspected Gilbert syndrome
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * creatinine ≤ institutional ULN OR
  * glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2 (see Appendix B).
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of relugolix and leuprolide on the developing human fetus are unknown. For this reason and because GnRH agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of relugolix or leuprolide depot administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of major adverse cardiac event, including myocardial infarction, new congestive heart failure (CHF) or CHF exacerbation, or stroke, within the past 6 months.
* Participants who have prior or planned concurrent treatment with second generation AR targeted therapies (such as abiraterone, enzalutamide, darolutamide, apalutamide).
* Participants who are receiving any other investigational agents.
* Patients with brain metastases will be excluded from the study as intermittent hormonal therapy is not standard of care treatment for this population.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to leuprolide depot or relugolix.
* Participants with uncontrolled intercurrent illness.
* Participant is unable to swallow pills.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
9-month Quality of Life (QOL) Score | At 9 months
  The QOL assessed using Functional Assessment of Cancer Therapy - Prostate (FACT-P) questionnaire, defined protocol section 11.1.1: The FACT-P (version 4) contains 39 Likert-type items distributed over 5 subscales: physical (7 items), social/family (7 items), emotional (6 items), and functional (7 items) well-being, and the additional concerns related to prostate cancer scale (12 items). The FACT-P total score is calculated by summing all these 5 subscales and ranges from 0 to 156.

SECONDARY OUTCOMES:
12-month Quality of Life (QOL) Score | At 12 months
  The QOL assessed using Functional Assessment of Cancer Therapy - Prostate (FACT-P) questionnaire, defined protocol section 11.1.1: The FACT-P (version 4) contains 39 Likert-type items distributed over 5 subscales: physical (7 items), social/family (7 items), emotional (6 items), and functional (7 items) well-being, and the additional concerns related to prostate cancer scale (12 items). The FACT-P total score is calculated by summing all these 5 subscales and ranges from 0 to 156.
9-month Hot flash related daily interference scale (HFRDIS) | At 9 months
  HFRDIS was Self-reported daily hot flash interference will be assessed with the Hot Flash-Related Daily Interference Scale, a valid and reliable measure used in prior prostate cancer studies. This scale assesses the impact of hot flashes on daily activities as well as overall quality of life. Total scores range from 0 - 100; higher scores indicate greater interference.
9-month Insomnia Severity Index (ISI) Score | At 9 months
  ISI Insomnia symptoms will be assessed using the ISI, which has been used in previous assessments of cancer patients, including men with prostate cancer. This questionnaire has 7 items asking about difficulties falling asleep, staying asleep, problems with waking too early and the satisfaction level with their current sleep pattern. Each item was rated on a scale from 0 to 4, where a higher score indicates a more severe insomnia.
9-month Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score | At 9 months
  Fatigue symptoms will be assessed with the FACIT-Fatigue survey, a valid and reliable instrument used in prostate cancer and other cancer studies, comprised of 13 items and rated on a 5 point Likert-type scale.
9-month EPIC-26 Sexual Function Summary Score | At 9 months
  Self-reported sexual function will be assessed using the sexual health section of the EPIC-26.
12-month Hot flash related daily interference scale (HFRDIS) | At 12 months
  HFRDIS was Self-reported daily hot flash interference will be assessed with the Hot Flash-Related Daily Interference Scale. This scale assesses the impact of hot flashes on daily activities as well as overall quality of life. Total scores range from 0 - 100; higher scores indicate greater interference.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Morgans, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Foxborough, Foxborough, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu